CLINICAL TRIAL: NCT04010461
Title: Theta Burst Transcranial Magnetic Stimulation of Fronto-parietal Networks: Modulation by Mental State
Acronym: TMScogMod
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephan F. Taylor, Professor of Psychiatry, University of Michigan
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HUM00165239; R21MH120633-01 (NIH)
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Results first posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: functional magnetic resonance imaging; Transcranial Magnetic Stimulation; dorsolateral prefrontal cortex

STUDY DESIGN:
Intervention Model Description: All participants will have 3 MRI sessions subsequent to the baseline visit and these will occur in a counterbalanced order.
Who Masked: Participant
Masking Description: All subjects will receive all interventions in a cross-over design. The three intervention sessions (visits 3, 4 & 5) will be given in counter-balanced order, stratified by gender. Subjects will be blind to the nature of the questions being asked; however, they will be told that different stimulation paradigms will be used, which will be evident to the subjects as they go through the procedures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- TMS to dlPFC, without a concurrent task (Experimental): TMS (intermittent theta burst stimulation) will be applied to the dlPFC, when subjects are in a resting state
  Interventions: Device: TMS; Behavioral: n-back working memory task
- TMS to vertex, without concurrent task (Experimental): TMS (intermittent theta burst stimulation) will be applied to the cerebral vertex, when subjects are in a resting state
  Interventions: Device: TMS; Behavioral: n-back working memory task
- TMS to dlPFC, during task (Experimental): TMS (intermittent theta burst stimulation) will be applied to the dlPFC, when subjects are engaged in the n-back working memory task
  Interventions: Device: TMS; Behavioral: n-back working memory task

INTERVENTIONS:
Device: TMS — Intermittent theta burst stimulation TMS applied to the cortex to excite cerebral cortex
  Other Names: intermittent theta burst stimulation (iTBS)
Behavioral: n-back working memory task — Subjects perform an executive function task, in which they view the serial presentation of letters and decide whether or not a letter matches a letter presented 'n' letters back (2 letters or 1 letter)

SUMMARY:
The purpose of this study is to improve understanding of the way transcranial magnetic stimulation (TMS), a form of non-invasive brain stimulation, affects the brain. The study hypothesis that when theta burst stimulation (TBS) is applied during a controlled mental state, network changes will be facilitated, compared to stimulation when mental state is uncontrolled. This study will focus on the dorsolateral prefrontal cortex (dlPFC) and the associated frontoparietal network (FPN), which subserves cognitive control - the ability to flexibly adapt and regulate behavior, an ability known to be impaired in neuropsychiatric conditions such as depression and dementia.

Healthy volunteers that qualify for this study will have psychological assessments and cognitive measures (due to Covid, some of these were done via teleconference), as well as functional Magnetic Resonance Imaging (fMRI) scans, completed after administration of TMS. Participants will be asked to come in for a total of five visits that include; a screening and assessment visit; a baseline functional magnetic resonance imaging (fMRI) scan, followed by TMS session; Visits 3, 4, and 5 will be the experimental TMS session, followed by fMRI scan.

DETAILED DESCRIPTION:
We will test the broad hypothesis that when TBS is applied during a controlled mental state, network changes will be facilitated, compared to stimulation when mental state is uncontrolled. We will focus on the dorsolateral prefrontal cortex (dlPFC) and the associated fronto-parietal network (FPN), which subserves cognitive control -- the ability to flexibly adapt and regulate behavior, an ability known to be impaired in neuropsychiatric conditions such as depression and dementia. We will use an 'n-back' task tapping cognitive control and the FPN. We will employ a within-subjects design with 40 healthy subjects in 4 MRI sessions. Each MRI session will consist of blood oxygenation level-dependent (BOLD) fMRI during an n-back task, resting state BOLD fMRI to measure connectivity and resting state arterial spin labeling (ASL) MRI to measure cerebral blood flow (rCBF) and examine effects on resting activity level. BOLD activation during the n-back will identify the FPN and the target site for dlPFC TBS. After a baseline fMRI session, subsequent sessions over different days will entail TBS, immediately followed by an MRI session to assess the effects of stimulation. TBS will involve: 1) dlPFC stimulation by active iTBS (600 pulses) alone or 2) while simultaneously performing an n-back cognitive task or 3) vertex (control) iTBS stimulation, alone.

ELIGIBILITY:
Inclusion Criteria:

* Women of child bearing age can not be pregnant or trying to become pregnant
* Ability to tolerate small, enclosed spaces without anxiety
* Size compatible with scanner gantry, e. g. men over 6 feet tall that weigh more than 250 lbs, men under 6 feet tall that weigh over 220 lbs, women over 5'11" tall that weigh more than 220 lbs, or women under 5'10" tall that weigh more than 200 lbs. Subjects of these weights or greater typically have difficult fitting into the fMRI scanner properly
* Ability and willingness to give informed consent to participate
* Alcohol or drug dependence (if in remission for greater than 5 years)

Exclusion Criteria

* History of past or current mental illness (except simple phobias)
* History of closed head injury, for example, loss of consciousness > approximately 5 minutes, hospitalization, neurological sequela;
* Metals, implants or metallic substances within or on the body that might cause adverse effects to the subject in a strong magnetic field, or interfere with image acquisition (for example; aneurysm clips, retained particles or metal workers with exposures, neurostimulators, foil-backed transdermal patches, carotid or cerebral stents, cerebral spinal fluid (CSF) shunts; magnetic dental implants, ferromagnetic ocular implants, pacemakers, and automatic implantable defibrillators).
* Prescription or non-prescription, with psychotropic effects (birth control medications allowed)
* First-degree family members with a history of epilepsy
* History of serious neurological illness or current medical condition that could compromise brain function, such as liver failure

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Taylor, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will share information about this/these trial(s) via timely registration, updates, and results reporting in ClinicalTrials.gov in accordance with NIH policy.
  The PI will also upload data gathered in this proposal to an National Institute of Mental Health (NIMH)-designated central data, NIMH Data Archive (NDA), as prescribed by NOT-MH-15-012, working with NIMH program to determine the timing and extent of data sharing. This includes formulation of an enrollment strategy that will obtain the information necessary to generate a Global Unique Identifier (GUID) for each participant.
  The consent form will include language indicating the intention to upload de-identified data into the central archive, and permission will be obtained from University of Michigan Institutional Review Board to do so. The budget includes a data manager to cover the costs of managing the data, building the data dictionary and harmonizing it with data structures.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified data will be entered into the NDA within 1 year of the conclusion of the study.
Access Criteria: No additional access restrictions will be placed on the de-identified data beyond those that are standard for the NDA.
URL: https://nda.nih.gov

REFERENCES:
- [Derived] Taylor SF, Lee TG, Jonides J, Tso IF, Hernandez-Garcia L. Theta Burst Transcranial Magnetic Stimulation of Fronto-Parietal Networks: Modulation by Mental State. J Psychiatr Brain Sci. 2020;5:e200011. doi: 10.20900/jpbs.20200011. Epub 2020 May 26. PMID 32613082

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 59 participants who were screened, 6 were ineligible and 53 were enrolled. With each treatment, regardless of the sequence, an MRI was performed.
Groups:
- All Groups: Since participants' data are only analyzed if they completed all assignments, and the order of assignment was immaterial to the trial, as it was a basic experiment studying humans, there was no reason to separate out the participants based on the order of interventions. Hence, the milestones listed below, other than "Completed," do not represent the actual sequential order for all participants.
Period: Overall Study
Arm/Group | All Groups
Started | 53
Participants Who Had Baseline Measurements | 47
TMS to dlPFC, Without a Concurrent Task (Passive) | 41
TMS to Vertex, Without Concurrent Task (Control) | 43
TMS to dlPFC, During Task (Active) | 40
Completed MRI Sessions | 40
Completed | 40
Not Completed | 13
Not completed — COVID based withdrawal | 5
Not completed — Withdrawal by Subject | 5
Not completed — Adverse Event | 1
Not completed — No Motor Threshold obtainable | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- All Groups: Since participants' data are only analyzed if they completed all assignments, and the order of assignment was immaterial to the trial, as it was a basic experiment studying humans, there was no reason to separate out the participants based on the order of interventions. Data is provided for all subjects whose data is analyzed.
Arm/Group | All Groups
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 24
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: 2-back Minus 1-back Blood Oxygen Level-Dependent (BOLD) Activation, Voxelwise in FPN
Description: Fronto-parietal network (FPN) defined by BOLD change while subject performed the n-back working memory task, contrasting high (2-back) versus low (1-back) loads. Using the SPM12 package, data were normalized per standard, open source routines. Using a General Linear Model framework, a model was estimated with regressors (after convolution with hemodynamic response function) for 2-back & 1-back conditions for each subject to predict BOLD change each day (arm).For analysis of group effects, second-level, between-subject analyses on normalized images of the 2-back minus 1-back beta estimate from the first level were entered into regression models, with mean frame displacement as a co-variate of no-interest to test contrasts between the arms/interventions. Using a FPN mask, the eigenvalues from the second-level estimates were extracted and entered into the analysis as an outcome measure. Note: eigenvalues are arbitrary units. Larger values indicate more BOLD signal.
Time Frame: 60 minutes after TMS during fMRI
Population: Of the 40 participants, image data from 3 failed quality control.
Measure: Mean (Standard Deviation); unit: arbitrary units
Groups:
- TMS to dlPFC, Without a Concurrent Task (Passive): TMS (intermittent theta burst stimulation) will be applied to the dlPFC, when subjects are in a resting state
  TMS: Intermittent theta burst stimulation TMS applied to the cortex to excite cerebral cortex
  n-back working memory task: Subjects perform an executive function task, in which they view the serial presentation of letters and decide whether or not a letter matches a letter presented 'n' letters back (2 letters or 1 letter)
- TMS to Vertex, Without Concurrent Task (Control): TMS (intermittent theta burst stimulation) will be applied to the cerebral vertex, when subjects are in a resting state
  TMS: Intermittent theta burst stimulation TMS applied to the cortex to excite cerebral cortex
  n-back working memory task: Subjects perform an executive function task, in which they view the serial presentation of letters and decide whether or not a letter matches a letter presented 'n' letters back (2 letters or 1 letter)
- TMS to dlPFC, During Task (Active): TMS (intermittent theta burst stimulation) will be applied to the dlPFC, when subjects are engaged in the n-back working memory task
  TMS: Intermittent theta burst stimulation TMS applied to the cortex to excite cerebral cortex
  n-back working memory task: Subjects perform an executive function task, in which they view the serial presentation of letters and decide whether or not a letter matches a letter presented 'n' letters back (2 letters or 1 letter)
Arm/Group | TMS to dlPFC, Without a Concurrent Task (Passive) | TMS to Vertex, Without Concurrent Task (Control) | TMS to dlPFC, During Task (Active)
Number analyzed (Participants) | 37 | 37 | 37
arbitrary units | 0.74 (0.54) | 0.75 (0.45) | 0.58 (0.39)
Statistical Analysis 1: Comparison: TMS to dlPFC, Without a Concurrent Task (Passive) vs TMS to dlPFC, During Task (Active); Analysis used standard, open-source methods for pre-processing . First-level analysis used the general framework of the modified General Linear Model, implemented in SPM12 with temporal convolution. For the n-back activation task, the first-level design matrix included regressors for 2-back and 1-back conditions, as well as 24 movement parameters. Statistical testing was done to establish whether more or less BOLD (neural activity) change occurred between two conditions; Test type: Superiority; p = 0.11, t-test, 2 sided; df = 35 Note: 1 subject was excluded from analysis as extraction of FPN eigenvalues failed due to technical deficiencies with image data; Mean Difference (Final Values) = 0.159, 95% CI 2-sided [-0.037 to 0.355], Standard Error of Mean 0.097
Statistical Analysis 2: Comparison: TMS to dlPFC, Without a Concurrent Task (Passive) vs TMS to Vertex, Without Concurrent Task (Control); Analysis used standard, open-source routes for slice timing correction, field map correction, realignment, smoothing (6 mm Gaussian kernel) and spatial normalization (MNI-152). First-level analysis used the general framework of the modified General Linear Model, implemented in SPM12 with temporal convolution. For the n-back activation task, the first-level design matrix included regressors for 2-back and 1-back conditions, as well as 24 movement parameters; Test type: Superiority; p = 0.94, t-test, 2 sided; df = 35 Note: 1 subject excluded from analysis as FPN extraction of eigenvalues failed due to technical issues with image data; Mean Difference (Final Values) = -0.009, 95% CI 2-sided [-0.245 to 0.227], Standard Error of Mean 0.116

2. Primary Outcome: Frontoparietal Network (FPN) Connectivity to Dorsolateral Prefrontal Cortex (dlPFC) Theta Burst Stimulation (TBS) Target
Description: Analysis of resting-state connectivity was performed used the CONN toolbox, using standard techniques to demonstrate connectivity between a spherical seed placed on each participant's locus of dlPFC stimulation, and the rest of the brain. Connectivity (correlations of BOLD signal) was first calculated for each participant, and then spatially averaged in MNI brain space, between participants. A 'cluster' of connectivity was identified, only if the number of voxels (thresholded at P <0.001) exceeded the count of 25. The outcome measure here is a count of the number of clusters exceeding this threshold, across all subjects. It represents significant connectivity between the site of stimulation and that cluster in the brain, for all subjects.
Time Frame: 60 minutes after TMS during fMRI
Population: 3 subjects failed image quality control processing
Measure: Number; unit: cluster count for connectivity
Arm/Group | TMS to dlPFC, Without a Concurrent Task (Passive) | TMS to Vertex, Without Concurrent Task (Control) | TMS to dlPFC, During Task (Active)
Number analyzed (Participants) | 37 | 37 | 37
cluster count for connectivity | 0 | 10 | 0
Statistical Analysis 1: Comparison: TMS to dlPFC, Without a Concurrent Task (Passive) vs TMS to dlPFC, During Task (Active); The contrast reflects the difference in connectivity between the conditions/sessions, at the level of each subject, then spatially averaged across all subjects. Functional connectivity strength for the dlPFC seed was represented by Fisher-transformed bivariate correlation coefficients from a weighted general linear model (weighted-GLM), defined separately for each pair of seed and target areas, modeling the association between their BOLD signal time series; Test type: Other — Group-level analyses were performed using a General Linear Model (GLM). For each individual voxel, a separate GLM was estimated, with first-level connectivity measures at this voxel as dependent variables, and groups or other subject-level identifiers as independent variables. Voxel-level hypotheses were evaluated using multivariate parametric statistics with random effects across subjects and sample covariance estimation across multiple measurements; p = 1, random field theory — Inferences were performed at the level of individual clusters (groups of contiguous voxels). Cluster-level inferences were based on parametric statistics from Gaussian Random Field theory; Results were thresholded using a combination of a cluster-forming p < 0.001 voxel-level threshold, and cluster-size threshold of 25 voxels; random field theory = 0 — Number indicates the number of clusters above the threshold of significance for the contrast between two arms (passive vs active)
Statistical Analysis 2: Comparison: TMS to dlPFC, Without a Concurrent Task (Passive) vs TMS to Vertex, Without Concurrent Task (Control); Results were thresholded using a combination of a cluster-forming p < 0.001 voxel-level threshold, and a corrected false discovery rate (FDR) p < 0.05 cluster-size threshold; Test type: Other — The applied test with random field theory uses a metric of spatial dispersion, testing against the null hypothesis that spatial clusters of difference across the analyzed region are no different from chance clustering; p = 1, random field theory; random field theory = 0 — Number indicates the number of clusters above the threshold of significance for the contrast between two arms (passive vs control)

3. Primary Outcome: Cerebral Blood Flow (rCBF) at Stimulation Target
Description: Regional cerebral blood flow measured at the site of theta burst stimulation (TBS) in milliliters per 100 mg tissue per minute
Time Frame: 15 minutes after TMS during fMRI
Population: pre-processing failures in 5 participants
Measure: Mean (Standard Deviation); unit: ml/100 mg tissue/min
Arm/Group | TMS to dlPFC, Without a Concurrent Task (Passive) | TMS to Vertex, Without Concurrent Task (Control) | TMS to dlPFC, During Task (Active)
Number analyzed (Participants) | 35 | 35 | 35
ml/100 mg tissue/min | 57.2 (20.7) | 57.9 (28.5) | 58.4 (20.3)
Statistical Analysis 1: Comparison: TMS to dlPFC, Without a Concurrent Task (Passive) vs TMS to Vertex, Without Concurrent Task (Control) vs TMS to dlPFC, During Task (Active); Test type: Superiority; p = 0.91, ANOVA; F-ratio = 0.10

4. Primary Outcome: Accuracy to 2-back
Description: Correct responses to letter stimuli, as a percentage of all responses
Time Frame: 60 minutes after TMS during fMRI
Population: Due to technical failures, data was lost for one participant during control and for 24 during "Active".
Measure: Mean (Standard Deviation); unit: percentage correct
Arm/Group | TMS to dlPFC, Without a Concurrent Task (Passive) | TMS to Vertex, Without Concurrent Task (Control) | TMS to dlPFC, During Task (Active)
Number analyzed (Participants) | 40 | 39 | 16
percentage correct | 96.7 (3.9) | 96.7 (3.6) | 96.2 (4.5)
Statistical Analysis 1: Comparison: TMS to dlPFC, Without a Concurrent Task (Passive) vs TMS to dlPFC, During Task (Active); Test type: Superiority; p = 0.55, ANOVA
Statistical Analysis 2: Comparison: TMS to dlPFC, Without a Concurrent Task (Passive) vs TMS to Vertex, Without Concurrent Task (Control); Test type: Superiority; p = .65, ANOVA

5. Secondary Outcome: 2-back Minus 1-back BOLD Activation, Voxelwise in Whole Brain
Description: Fronto-parietal network (FPN) defined by BOLD change while subject performed the n-back working memory task, contrasting high (2-back) versus low (1-back) loads. Using the SPM12 package, data were normalized per standard, open source routines. Using a General Linear Model framework, a model was estimated with regressors (after convolution with hemodynamic response function) for 2-back & 1-back conditions for each subject to predict BOLD change each day (arm).For analysis of group effects, second-level, between-subject analyses on normalized images of the 2-back minus 1-back beta estimate from the first level were entered into regression models. With a cluster threshold of voxel magnitude < 0.001, clusters of difference are defined. Because there are often multiple clusters in a contrast, the number below is the size, in voxels, of the largest cluster, across all participants, for each session.
Time Frame: 60 minutes after TMS during fMRI
Population: 3 participants were not analyzed due to poor data quality
Measure: Number; unit: voxel count
Arm/Group | TMS to dlPFC, Without a Concurrent Task (Passive) | TMS to Vertex, Without Concurrent Task (Control) | TMS to dlPFC, During Task (Active)
Number analyzed (Participants) | 37 | 37 | 37
voxel count | 1139 | 1532 | 907
Statistical Analysis 1: Comparison: TMS to dlPFC, Without a Concurrent Task (Passive) vs TMS to dlPFC, During Task (Active); Statistical thresholding using a random field model adjusted for multiple comparisons, with initial voxel magnitude/height threshold set at p < 0.001 and peak and cluster-corrected significance levels obtained (false discovery rate [FDR]corrected), across the entire brain; Test type: Other; p = 0.54, random field theory — P-value above represents the lowest (most significant) value of the largest cluster, for the contrast of Passive > Active, testing whether the cluster size is greater than chance; cluster size = 42 — The estimated parameter is the size, in voxels, of the largest cluster. The applied test with random field theory tests whether the size of cluster difference across are no different from chance clustering
Statistical Analysis 2: Comparison: TMS to dlPFC, Without a Concurrent Task (Passive) vs TMS to Vertex, Without Concurrent Task (Control); [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.93, random field theory — P-value above represents the lowest (most significant) value of the largest cluster, for the contrast of Passive > Control, testing whether the size of this cluster is greater than one would expect by chance alone; cluster size = 16 — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Measure Cerebral Blood Flow (rCBF) in FPN
Description: Regional cerebral blood flow measured in the FPN in milliliters per 100 mg tissue per minute
Time Frame: 15 minutes after TMS during fMRI
Population: 5 subjects with poor data quality had to be excluded
Measure: Mean (Standard Deviation); unit: mL/100 mg tissue/min
Arm/Group | TMS to dlPFC, Without a Concurrent Task (Passive) | TMS to Vertex, Without Concurrent Task (Control) | TMS to dlPFC, During Task (Active)
Number analyzed (Participants) | 35 | 35 | 35
mL/100 mg tissue/min | 52.7 (11.8) | 52.9 (15.6) | 51.9 (13.1)
Statistical Analysis 1: Comparison: TMS to dlPFC, Without a Concurrent Task (Passive) vs TMS to Vertex, Without Concurrent Task (Control) vs TMS to dlPFC, During Task (Active); Repeated measures ANOVA to test for differences in cerebral blood flow (perfusion) in the frontoparietal network; Test type: Superiority; p = 0.8, ANOVA; F-ratio = 0.22

7. Secondary Outcome: Median Reaction Time (RT) in 2-back
Description: Median reaction time for subjects responding in the n-back task, for correct responses (1-back and 2-back)
Time Frame: 60 minutes after TMS during fMRI
Population: Due to technical failures, data was lost for one participant during control and for 24 participants during "Active".
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | TMS to dlPFC, Without a Concurrent Task (Passive) | TMS to Vertex, Without Concurrent Task (Control) | TMS to dlPFC, During Task (Active)
Number analyzed (Participants) | 40 | 39 | 16
milliseconds | 573.2 (175.8) | 556.4 (164.2) | 572.1 (135.4)
Statistical Analysis 1: Comparison: TMS to dlPFC, Without a Concurrent Task (Passive) vs TMS to dlPFC, During Task (Active); Test type: Superiority; p = 0.06, ANOVA; F-ratio = 3.96
Statistical Analysis 2: Comparison: TMS to dlPFC, Without a Concurrent Task (Passive) vs TMS to Vertex, Without Concurrent Task (Control); Test type: Superiority; p = 0.68, ANOVA; F-ratio = 0.17

8. Secondary Outcome: D-prime in 2-back
Description: d-prime = z(H) - z(F) , where z(H) and z(F) are the z transforms of hit rate and false alarm, respectively.
  Hit rate = number of correctly identified targets/number of targets presented False alarm = number of incorrectly identified targets/number of non-targets presented
Time Frame: 60 minutes after TMS during fMRI
Population: Due to technical failures, data was lost for one participant during control and for 24 participants during "Active".
Measure: Mean (Standard Deviation); unit: d-prime
Arm/Group | TMS to dlPFC, Without a Concurrent Task (Passive) | TMS to Vertex, Without Concurrent Task (Control) | TMS to dlPFC, During Task (Active)
Number analyzed (Participants) | 40 | 39 | 16
d-prime | 3.8 (0.7) | 3.8 (0.6) | 3.7 (0.8)
Statistical Analysis 1: Comparison: TMS to dlPFC, Without a Concurrent Task (Passive) vs TMS to dlPFC, During Task (Active); Test type: Superiority — Repeated measures ANOVA for 1- and 2-back conditions; p = 0.41, ANOVA; F-ratio = 0.72
Statistical Analysis 2: Comparison: TMS to dlPFC, Without a Concurrent Task (Passive) vs TMS to Vertex, Without Concurrent Task (Control); Test type: Superiority; p = 0.50, ANOVA

ADVERSE EVENTS:
Time Frame: duration of participation in study -- 3- 6 weeks
Groups:
- Baseline Measurement: Initial assessments, baseline MRI scan, TMS motor threshold
Arm/Group | Baseline Measurement | TMS to dlPFC, Without a Concurrent Task (Passive) | TMS to Vertex, Without Concurrent Task (Control) | TMS to dlPFC, During Task (Active)
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/41 | 0/43 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/41 | 0/43 | 0/40
Other Adverse Events (participants affected / at risk) | 4/47 | 2/41 | 0/43 | 1/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline Measurement (N=47) | TMS to dlPFC, Without a Concurrent Task (Passive) (N=41) | TMS to Vertex, Without Concurrent Task (Control) (N=43) | TMS to dlPFC, During Task (Active) (N=40)
Finger/Hand Soreness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 | 0 | 0
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 | 0
Lightheadedness (Nervous system disorders) | 0 | 1 (1) | 0 | 0
Discomfort During fMRI (General disorders) | 1 (1) | 0 | 0 | 1 (1)

LIMITATIONS AND CAVEATS:
Because of technical problems, performance measure for accuracy and d-prime were not available for 24 subjects in the 'Active' condition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT04010461/Prot_SAP_002.pdf
  • Informed Consent Form (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/61/NCT04010461/ICF_000.pdf